CLINICAL TRIAL: NCT02837081
Title: The Impact of Preauthorization Compared to Prospective Audit on Outcome Indicators as Core Strategies of Antimicrobial Stewardship Program
Brief Title: Preauthorization Versus Prospective Audit in Antimicrobial Stewardship Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Susan Shin-Jung Lee, Attending physician, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VGHKS15-CT12-05
Record Dates: First submitted 2015-12-01; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preauthorization group (Active Comparator): Strategy 1 of antimicrobial stewardship: Prescriptions of antimicrobial agents are done real-time by infectious diseases physician consultant. Use restricted without real-time authorization.
  Interventions: Other: preauthorization strategy of antimicrobial stewardship
- Prospective audit (Experimental): Strategy 2 of antimicrobial stewardship: Prescription of antimicrobial agents are audited 48-72 hours later by infectious diseases physician consultant. Use allowed without authorization for 72 hours.
  Interventions: Other: Prospective audit strategy of antimicrobial stewardship

INTERVENTIONS:
Other: Prospective audit strategy of antimicrobial stewardship — applying prospective audit as a different strategy of antimicrobial stewardship
  Other Names: prospective audit
  Arms: Prospective audit
Other: preauthorization strategy of antimicrobial stewardship — applying preauthorization as one strategy of antimicrobial stewardship
  Other Names: preauthorization
  Arms: Preauthorization group

SUMMARY:
Antimicrobial stewardship program (ASP) is recommended to improve appropriate antimicrobial use, reduce bacterial resistance, unnecessary drug costs and enhance patient health outcomes. Two core strategies of ASP recommended as effective in guidelines are formulary restriction with drug preauthorization and prospective audit with feedback. Investigators will evaluate the effectiveness of the 2 strategies using antimicrobial utilization and patient outcomes.

DETAILED DESCRIPTION:
Background: Antimicrobial stewardship program (ASP) is recommended to improve appropriate antimicrobial use, reduce bacterial resistance, unnecessary drug costs and enhance patient health outcomes. Two core strategies of ASP recommended as effective in guidelines are formulary restriction with drug preauthorization and prospective audit with feedback. Preauthorization is the current strategy used in our hospital, while most other hospitals in Taiwan and worldwide uses prospective audit with feedback. Preauthorization requires intensive manpower to maintain timeliness of antimicrobial use. This study will evaluate a policy change in strategy used for antimicrobial stewardship. Investigators will evaluate the effectiveness of the 2 strategies using antimicrobial utilization and patient outcomes.

Methods: During a stepwise change in the policy of the antimicrobial stewardship program in this hospital, the study will observe the differences between two standardized core strategies (preauthorization vs prospective audit) of ASP. Hospitalized patients aged 20 and above, requiring use of restricted antimicrobials will be recruited into the study. Signing of consent forms are waived since both strategies are already proven to be effective and are widely implemented in Taiwan and worldwide. Also, the evaluation of such policy changes will not impact on patient safety or patient rights. The conduction of the study will not require contacting patients and no clinical samples will be collected. All data required for analysis will be collected via a computerized patient care system. Patient data will be protected via de-linking. Patients will be excluded if admitted at or entered the intensive care unit within 48 hours of entry, and if infectious diseases consultation had been requested. Eligible patients will be randomized to either preauthorization, which is the current practice in the hospital; or prospective audit, that will be done at 48-72 hours after prescription, as is the current practice in other hospitals in Taiwan and worldwide. Managing physicians are not obligated to follow our advice and the investigators will not intervene in their management decisions. Primary outcomes include antimicrobial utilization, drug costs and patient outcomes such as length of stay and clinical improvement. The time spent on implementing these two strategies will be compared.

The study hypothesis is that the preauthorization group will impact on a reduction in antimicrobial cost and utilization, especially in the first 72 hours, when compared to prospective audit. However, patient outcomes will likely be similar. Antimicrobial stewardship programs using preauthorization as a core strategy compared to prospective audit with feedback have similar patient outcomes, but may reduce antimicrobial utilization.

ELIGIBILITY:
Inclusion Criteria:

* In-hospital patients, aged 20 and above, with request from managing physicians for use of restricted antimicrobials.

Exclusion Criteria:

* Patients admitted to the intensive care unit at evaluation or within 48 hours of entry into the study.
* Patients with antimicrobial prescriptions prescribed during after-hours, including weekends and public holidays.
* Formal infectious disease consultations requested prior to randomization.
* Patients in the emergency department and outpatient department.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Antimicrobial utilization using defined daily dose (DDD) | 4 weeks
  Defined daily dose (DDD),
Antimicrobial utilization using defined daily dose per 1000 patient days (DID) | 4 weeks
  Defined daily dose per 1000 patient days

SECONDARY OUTCOMES:
Appropriateness of antimicrobial prescription by susceptibility of culture | 4 weeks
  cultures shows susceptibility to antimicrobial prescribed
Rate of acceptance to use antimicrobial agents recommended by infectious disease physicians | 4 weeks
  choice of antimicrobial agents used matches recommendation by infectious diseases physician

OTHER OUTCOMES:
30-day mortality | 30 days post randomization
  mortality rate at 30-days post randomization
3-day defervescence rate | 3 day post randomization
  Rate of defervescence on day 3 post randomization
Rate of hospital associated bloodstream infections | 12 months
  overall rate of bloodstream infection within the hospital during the study period
Rates of multidrug resistant organisms within the hospital | 12 months
  Rates of carbapenem-resistant Acinetobacter baumanii (CRAB), vancomycin resistant Enterococcus (VRE), Clostridium difficile

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shin-Jung Lee, M.D., Ph.D., Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Society for Healthcare Epidemiology of America; Infectious Diseases Society of America; Pediatric Infectious Diseases Society. Policy statement on antimicrobial stewardship by the Society for Healthcare Epidemiology of America (SHEA), the Infectious Diseases Society of America (IDSA), and the Pediatric Infectious Diseases Society (PIDS). Infect Control Hosp Epidemiol. 2012 Apr;33(4):322-7. doi: 10.1086/665010. PMID 22418625
- [Result] W.H.O. (2011) WHO Global Strategy for Containment of Antimicrobial Resistance.
- [Result] Tseng SH, Lee CM, Lin TY, Chang SC, Chuang YC, Yen MY, Hwang KP, Leu HS, Yen CC, Chang FY. Combating antimicrobial resistance: antimicrobial stewardship program in Taiwan. J Microbiol Immunol Infect. 2012 Apr;45(2):79-89. doi: 10.1016/j.jmii.2012.03.007. Epub 2012 Apr 5. PMID 22483434
- [Result] Dellit TH, Owens RC, McGowan JE Jr, Gerding DN, Weinstein RA, Burke JP, Huskins WC, Paterson DL, Fishman NO, Carpenter CF, Brennan PJ, Billeter M, Hooton TM; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America. Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America guidelines for developing an institutional program to enhance antimicrobial stewardship. Clin Infect Dis. 2007 Jan 15;44(2):159-77. doi: 10.1086/510393. Epub 2006 Dec 13. No abstract available. PMID 17173212
- [Result] Chung GW, Wu JE, Yeo CL, Chan D, Hsu LY. Antimicrobial stewardship: a review of prospective audit and feedback systems and an objective evaluation of outcomes. Virulence. 2013 Feb 15;4(2):151-7. doi: 10.4161/viru.21626. Epub 2013 Jan 9. PMID 23302793
- [Result] Lin YS, Lin IF, Yen YF, Lin PC, Shiu YC, Hu HY, Yang YP. Impact of an antimicrobial stewardship program with multidisciplinary cooperation in a community public teaching hospital in Taiwan. Am J Infect Control. 2013 Nov;41(11):1069-72. doi: 10.1016/j.ajic.2013.04.004. Epub 2013 Jul 17. PMID 23870295
- [Result] Teng CB, Ng TM, Tan MW, Tan SH, Tay M, Lim SF, Ling LM, Ang BS, Lye DC. Safety and effectiveness of improving carbapenem use via prospective review and feedback in a multidisciplinary antimicrobial stewardship programme. Ann Acad Med Singap. 2015 Jan;44(1):19-25. PMID 25703493
- [Result] Reed EE, Stevenson KB, West JE, Bauer KA, Goff DA. Impact of formulary restriction with prior authorization by an antimicrobial stewardship program. Virulence. 2013 Feb 15;4(2):158-62. doi: 10.4161/viru.21657. Epub 2012 Nov 15. PMID 23154323
- [Result] Mehta JM, Haynes K, Wileyto EP, Gerber JS, Timko DR, Morgan SC, Binkley S, Fishman NO, Lautenbach E, Zaoutis T; Centers for Disease Control and Prevention Epicenter Program. Comparison of prior authorization and prospective audit with feedback for antimicrobial stewardship. Infect Control Hosp Epidemiol. 2014 Sep;35(9):1092-9. doi: 10.1086/677624. Epub 2014 Jul 23. PMID 25111916
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] W.H.O. Defined Daily Dose (DDD). 2015 [cited 2015 May 24]; Available from: http://www.whocc.no/ddd/definition_and_general_considera/.
- [Result] van den Bosch CM, Geerlings SE, Natsch S, Prins JM, Hulscher ME. Quality indicators to measure appropriate antibiotic use in hospitalized adults. Clin Infect Dis. 2015 Jan 15;60(2):281-91. doi: 10.1093/cid/ciu747. Epub 2014 Sep 28. PMID 25266285